CLINICAL TRIAL: NCT04983134
Title: Women Helping Women Lung Cancer Screening (WHW-L)
Brief Title: Women Helping Women - Lung Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OCR40152; IRB202100009 (Other: University of Florida)
Record Dates: First submitted 2021-06-30; First posted 2021-07-30 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Intervention(SI) (No Intervention): the HealthStreet Standard Intervention to include a CHW referral to an accessible and acceptable lung cancer screening site to include a financial counselor (if needed), tobacco cessation and quit resources (if still smoking) and, additionally, will watch the Genentech lung cancer screening video with the CHW;
- Enhanced CHW Intervention (Experimental): After 1:1 randomization, 30 women will additionally receive a 6-hour four week Enhanced CHW Intervention (E-CHW-I) modelled on successful peer-partnered interventions and informed by Stages of Change theory, which will add to the SI, calls and texts (if appropriate) to help problem solve and encourage screening receipt and transportation to the screening (if needed);
  Interventions: Behavioral: Enhanced CHW Intervention

INTERVENTIONS:
Behavioral: Enhanced CHW Intervention — community-based intervention
  Arms: Enhanced CHW Intervention

SUMMARY:
The Women Helping Women Lung Cancer Screening (WHW-L) Study will be conducted to develop a scalable, easy to apply community-based intervention to increase rates of lung cancer screening and follow-up in high-need/low-resource populations, based on a Transtheoretical Stages of Change theoretical model. The investigators will test the feasibility of using Community Health Workers to recruit (Aim 1) and partner with 60 community members (Aim 2) within 6 months, to take the steps to consult with a doctor, schedule screening, and/or attend screening (Aim 3) [84 people may be screened for the study assuming some don't continue}.CHWs will use the HealthStreet 12,000+ cohort to identify current or former female smokers (adults 50 to 77 years old) with a smoking history of 25 pack-years who could benefit from LDCT screening for lung cancer and will facilitate steps in their screening receipt. All participants will benefit from the Standard Intervention; additionally, a random sample of 30 will receive the Enhanced CHW Intervention (E-CHW-I). The investigators hypothesize that women who may be at higher risk of lung cancer due to lack of knowledge, access, and resources will take steps to receipt of LDCT in both interventions, with those receiving the Enhanced Intervention more likely to take these steps. Ultimately, such an intervention could lead to a lower lung cancer burden in the target population

ELIGIBILITY:
Inclusion Criteria:

* women who are 50 to 80 years old
* 20+ pack-years of smoking history
* live within 45 miles of UF Health Shands Hospital or in Duval County, specifically the 12,000+ HealthStreet cohort

Exclusion Criteria:

* women outside the acceptable age range
* insufficient smoking history
* women who live outside the 45 miles of UF Health Shands Hosptial or not in Duval County not in the HealthStreet system

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Feasibility of Recruitment - Degree of Agreement Measured with Likert Scale | at baseline visit
  Feasibility of recruiting occurs with the Baseline Assessment which will assess participants' degree of agreement with their readiness to receive lung cancer screening on a 10 point Likert scale (strongly disagree through strongly agree) mirroring those used to assess readiness for breast and colorectal cancer screening
Feasibility of Implementation - screening adherence with Community Health Worker | At 4 weeks after intervention completion
  to test the feasibility of implementation of a customize culturally relevant, gender-specific Community Health Worker partnered intervention using the Transtheoretical Stages of Change model, the investigators will measure screening adherence in hours for lung cancer among the 60 women assessed through records of intervention delivery, including Randomization and Contact Logs, where the investigators will document each contact with the 60 women enrolled.
Evaluation of Efficacy - number of participants who engaged in a referred screening service | after intervention completion, at the 45-day follow up call
  to evaluate the limited efficacy of the WHW-L intervention to increase screening for lung cancer among the 60 women at 45 days to improve outcome variables: see physician re lung cancer screening/smoking, schedule screening, receive screening, the investigators will conduct phone-based follow-up interviews among all 60 women at 45 days.

CONTACTS AND LOCATIONS:
Locations (1):
- UF Health Cancer Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No